CLINICAL TRIAL: NCT06313398
Title: Determination of Red Cell Survival in Sickle Cell Disease and Other Hemoglobinopathies Using Biotin Labeling
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10001883; 001883-H
Record Dates: First submitted 2024-03-14; First posted 2024-03-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Sickle Cell Disease; Thalassemia; Hemoglobinopathy
Keywords: Red Cell; Hemoglobinopathy; Thalassemia; Sickle Cell Disease; Biotin
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Hemoglobinopathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RBC survival in patients with SCD (Experimental): RBC lifespan, determined by the mean number of days from biotin-labeled RBC infusion until biotin-labeled RBCs are below limit of detection, in patients with inherited hemoglobinopathies prior to and post initiation of disease modifying therapy or HSCT
  Interventions: Biological: Biotin-labeled red blood cells

INTERVENTIONS:
Biological: Biotin-labeled red blood cells — Cellular Product (patient's own red blood cells washed in Biotin and infused back to patient)

SUMMARY:
Background:

Sickle cell disease (SCD) is an inherited disorder of the blood. SCD causes red blood cells (RBCs) to die early. This can lead to a shortage of healthy cells. SCD and other blood disorders can be managed with drugs or cured with a bone marrow transplant. Researchers want to know how long RBCs survive in people with SCD and other blood disorders before and after treatment compared to those who had a bone marrow transplant.

Objective:

To learn how long RBCs survive in the body in people with SCD and other blood disorders compared to those whose disease was cured with a bone marrow transplant.

Eligibility:

People aged 18 years or older with SCD or another inherited blood disorder. People whose SCD or blood disorder was cured with a bone marrow transplant are also needed.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests.

Participants will have about 7 tablespoons of blood drawn. In the lab, this blood will be mixed with a vitamin called biotin. Biotin sticks to the outside of RBCs. This process is called "biotin labeling of RBCs." The next day, the participant s own biotin-labeled RBCs will be returned to their bloodstream.

Participants will return regularly to have smaller blood samples (about 2 teaspoons) drawn. These samples will be tested to detect the percentage of cells that have biotin labels. These visits may be every 2 weeks, 4 weeks, or some other interval. Participants will continue this schedule for up to 20 weeks or until biotin can no longer be detected....

DETAILED DESCRIPTION:
Study Description:

This study will use biotin-labeling of red blood cells (RBCs) to determine the mean potential lifespan (MPL) of RBCs in patients with sickle cell disease (SCD) and other hemoglobinopathies (e.g. thalassemia), including in those receiving disease modifying therapies or who have undergone curative hematopoietic stem cell transplantation (HSCT: allogeneic or autologous). Previous studies have corroborated the MPL of healthy donor RBCs to be approximately 115 days, while RBCs from patients with SCD have a more variable but consistently shorter MPL of approximately 32 days. We recently validated these findings and demonstrated the feasibility, safety, and efficacy of determining MPL of biotin-labeled RBCs in patients with SCD before and after transplant, persons with sickle cell trait, and healthy donors. Allogeneic HSCT is a curative treatment for severe SCD with stable, mixed donor-recipient chimerism after HSCT sufficient to reverse the sickle cell phenotype by virtue of improved donor red cell survival compared to the ineffective erythropoiesis of SCD. HSCT, both allogeneic and autologous, are also curative for certain hemoglobinopathies, such as transfusion dependent beta thalassemia (TDT), with donor cells able to overcome the ineffective erythropoiesis in TDT as well. We predict that the hematologic variables associated with red cell survival among patients with SCD and other hemoglobinopathies vary between individuals and are affected by disease modifying therapy, including curative therapies. The data generated will refine our understanding of the degree of correction necessary to reverse the clinical phenotype of SCD and other hemoglobinopathies, including that needed for autologous gene therapy to be curative.

Objectives:

Primary Objective:

To determine and compare red blood cell survival, by virtue of the mean number of days of detectable biotin-labeled RBCs, in participants with SCD and/or other hemoglobinopathies before and after initiation of disease modifying therapy, including those who have undergone HSCT.

Secondary Objective:

To validate the association of red cell survival with known markers of increased survival, specifically absolute reticulocyte count, hemoglobin F or hemoglobin A percentage, and alpha globin mutation status (SCD participants only).

Exploratory Objective:

To create and pilot a mathematical model incorporating RBC survival and reticulocyte count to determine the necessary amount of normal hemoglobin or hemoglobin F needed to reverse sickle cell complications. Information from participants with inherited high HbF will be used.

Endpoints:

Primary Endpoint:

Red blood cell survival via measurement of detectable biotin-labeled RBC with time

Secondary Endpoint:

Relationship of RBC survival to hematologic parameters.

Exploratory Endpoint:

Amount of normal hemoglobin or hemoglobin F needed to reverse the sickle cell complications.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or greater with confirmed diagnosis of SCD (all genotypes), thalassemia (beta and/or alpha), or other inherited hemoglobinopathy not otherwise specified.
4. Be at steady state for their underlying disease (e.g. SCD or thalassemia) or post-bone marrow transplantation status, as evidenced by medical history.
5. Ability to have blood samples drawn.
6. For female participants of child-bearing potential, agree to use birth control during study participation. Female subjects of child-bearing potential must agree to use a medically acceptable method of birth control such as an oral contraceptive, intrauterine device, barrier and spermicide, or contraceptive implant/injection from start of screening through 4 months after infusion.
7. Agreement to adhere to Lifestyle Considerations throughout study duration

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Consumption of biotin supplements or raw eggs within the last 30 days.
2. Blood loss within the previous 8 weeks (>540 mL).
3. Red cell transfusion for their underlying SCD and/or thalassemia within the last 3 months.

   a. Participants may be eligible after three months following their last transfusion.
4. Patients on hemodialysis, due to possibility of early removal of biotinylated RBCs.
5. Pregnancy, lactation or absence of adequate contraception for fertile female subjects.
6. Pediatric subjects will not participate in this study.
7. Known allergic reactions to biotin, due to risk of possible life-threatening allergic reaction.
8. Current diagnosis of malignancy (liquid and/or solid).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
To determine and compare red blood cell survival, by virtue of the mean number of days of detectable biotin-labeled RBCs, in participants with SCD and/or other hemoglobinopathies. | Patients w/o transplant: lab draw every 2 weeks until biotin-labeled cells are no longer detected. Patients Post-transplant: lab draw every four weeks, until week 12. Lab draw every 2 weeks until biotin-labeled cells are no longer detected.
  Enumeration of biotin-labeled RBCS (BioRBCs) will be performed by flow cytometry. F-cell and/or S-cell measurement will be done by flow cytometry. BioRBCs will be isolated from post-infusion blood samples using flow cytometry separation. The collected BioRBCs and the whole blood fraction will be analyzed by high performance liquid chromatography (HPLC) for hemoglobin content.

SECONDARY OUTCOMES:
Validate the association of RBC survival with known markers of increased survival. | Patients w/o transplant: lab draw every 2 weeks until biotin-labeled cells are no longer detected. Patients Post-transplant: lab draw every four weeks, until week 12. Lab draw every 2 weeks until biotin-labeled cells are no longer detected.
  We will measure the relationship of RBC survival to hematologic parameters known to be associated with survival, specifically hemolysis markers (e.g. absolute reticulocyte count, lactate dehydrogenase, total bilirubin, and aspartate aminotransferase), hemoglobin F or hemoglobin A percentage, and alpha globin gene mutation status obtained at baseline and during scheduled lab draws (except for alpha globin gene mutation analysis which is only done at baseline).

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001883-H.html